CLINICAL TRIAL: NCT01781754
Title: Changes in UCP2 mRNA in T2DM Patients
Brief Title: Changes in Mitochondrial Uncoupling Protein 2 (UCP2) Messenger RNA(mRNA) in Type 2 Diabetes (T2DM) Patients
Acronym: Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-11-NV-561-CTIL
Record Dates: First submitted 2013-01-08; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes
Keywords: Glycemic control; Metabolic control; Oxidative stress; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood for UCP2 mRNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic patients: Un balanced diabetic patients
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — This is the only intervention that is part of the study. A family physician or other physician will be responsible of the diabetic treatment (common treatment, e.g Metformin).

SUMMARY:
Many patients with Diabetes find difficulties in achieving glycemic control. Hemoglobin A1c(HgBA1c) is used as a marker for glycemic control. UCP2 is affected by high glucose levels, high free fatty acids and high oxidative stress.

The investigators intend to learn about the changes in UCP2 along the process of reaching glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Un balanced diabetic patients.

Exclusion Criteria:

* No current infection.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Un balanced diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Levels of gene expression for UCP2 (RQ) | 6 months
  Checking UCP2 levels compared to HgBA1c

SECONDARY OUTCOMES:
Improved metabolic state | 6 months
  Glycemic control (glucose level and HgA1c), levels of free reactive oxygen species (ROS) and non-esterified fatty acids (NEFAs).

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Dmitriev AD, Factor MI, Segal OL, Pavlova EV, Massino YS, Smirnova MB, Yakovleva DA, Dmitriev DA, Kizim EA, Kolyaskina GI, Brusov OS. Western blot analysis of human and rat serotonin transporter in platelets and brain using site-specific antibodies: evidence that transporter undergoes endoproteolytic cleavage. Clin Chim Acta. 2005 Jun;356(1-2):76-94. doi: 10.1016/j.cccn.2004.12.019. Epub 2005 Mar 17. PMID 15936305
- [Background] Rudofsky G Jr, Schroedter A, Schlotterer A, Voron'ko OE, Schlimme M, Tafel J, Isermann BH, Humpert PM, Morcos M, Bierhaus A, Nawroth PP, Hamann A. Functional polymorphisms of UCP2 and UCP3 are associated with a reduced prevalence of diabetic neuropathy in patients with type 1 diabetes. Diabetes Care. 2006 Jan;29(1):89-94. doi: 10.2337/diacare.29.01.06.dc05-0757. PMID 16373902
- [Background] Dulloo AG, Samec S. Uncoupling proteins: their roles in adaptive thermogenesis and substrate metabolism reconsidered. Br J Nutr. 2001 Aug;86(2):123-39. doi: 10.1079/bjn2001412. PMID 11502224
- [Background] Schrauwen P, Hesselink M. UCP2 and UCP3 in muscle controlling body metabolism. J Exp Biol. 2002 Aug;205(Pt 15):2275-85. doi: 10.1242/jeb.205.15.2275. PMID 12110661
- [Background] Rendel M. Advances in diabetes for the millennium: nutritional therapy of type 2 diabetes. MedGenMed. 2004 Sep 1;6(3 Suppl):10. PMID 15647715
- [Background] Krauss S, Zhang CY, Lowell BB. The mitochondrial uncoupling-protein homologues. Nat Rev Mol Cell Biol. 2005 Mar;6(3):248-61. doi: 10.1038/nrm1592. PMID 15738989
- [Background] Borecky J, Vercesi AE. Plant uncoupling mitochondrial protein and alternative oxidase: energy metabolism and stress. Biosci Rep. 2005 Jun-Aug;25(3-4):271-86. doi: 10.1007/s10540-005-2889-2. PMID 16283557